CLINICAL TRIAL: NCT05194371
Title: Report of the Survival Outcomes of Patients With Esophageal Cancer After Definitive Radiotherapy in China
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: YW2021-92-1
Record Dates: First submitted 2021-12-24; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Definitive (chemo)radiotherapy
  Interventions: Radiation: definitive radiotherapy or definitive chemoradiotherapy

INTERVENTIONS:
Radiation: definitive radiotherapy or definitive chemoradiotherapy — A total dose of radiation therapy should be more than 50Gy

SUMMARY:
In this study, data of esophageal cancer patients undergoing definitive radiotherapy in 14 institutions from various provinces in China were evaluated to help strengthen confidence in anti-cancer, including rehabilitation, economic burden, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with esophageal cancer who received definitive radiotherapy (radiotherapy dose ≥50Gy) from 2015 to 2016
2. Age ≥ 18
3. The radiation field included primary esophageal tumor with or without lymph node metastasis

Exclusion Criteria:

1. Radiotherapy dose < 50Gy
2. Palliative radiotherapy
3. The radiation field are metastatic areas, such as bone, brain, adrenal gland, isolated metastatic lymph nodes, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer who received definitive radiotherapy (radiotherapy dose ≥50Gy) from 2015 to 2016 in 14 institutions in China
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 year

SECONDARY OUTCOMES:
the European Organisation for Research and Treatment of Cancer (EORTC) questionnaire module to assess quality of life (QOL) | 5 year
  The EORTC QLQ-core 30 questionnaire is composed of multi-item scales and single-item measures including 5 functional scales, 3 symptom scales, a global health status-QoL scale, and 6 single items. Each of the multi-item scales includes a different set of items - no item occurs in more than 1 scale. High scale score=higher response level; a high score for a functional scale=a healthy level of function, high score for the global health status/QoL=high quality of life but a high score for a symptom scale / item=high level of symptomatology/problems. The principle for scoring these scales: 1.) Estimate the average of the items that contribute to the scale = raw score. 2.) Linear transformation to standardize the raw score, so that scores range from 0 to 100. Results should be interpreted with caution as the numbers of patients with available data over time were limited, and because of high variances as evidenced by large standard deviations.
Costs of treatment | 5 year
  Financial burden, Whether medical insurance is affordable
Proportion of using chemotherapy or target therapy concurrently with radiotherapy | 2 month
  Medication

CONTACTS AND LOCATIONS:
Overall Officials: Lvhua Wang, Principal Investigator — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital, Chinese Academy of Medical Sciences and Peking Union Medic; Kuaile Zhao, Principal Investigator — Fudan University
Locations (1):
- Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China